CLINICAL TRIAL: NCT00015561
Title: Pesticides--Health Fertility and Reproductive Risk
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 8161-CP-001
Record Dates: First submitted 2001-04-20; First posted 2001-04-23 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Birth Defects; Miscarriages; Cancer
Keywords: population studies; laboratory evaluation; hormone analysis; semen analysis; chromosome studies
MeSH Terms: conditions — Congenital Abnormalities; Abortion, Spontaneous; Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This project is designed to establish whether pesticides or other environmental agents have a role in the excess birth defects identified in the Red River Valley of Minnesota. In this human study, laboratory based health parameters will be used to key in health survey data. In vitro data will be developed to mechanistic information. Concordant results among these study features will provide a weight of evidence approach.

ELIGIBILITY:
Pesticide applicators and their spouses

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1803
Dates: Start 1996-09; Study Completion 2001-08

CONTACTS AND LOCATIONS:
Overall Officials: Vincent F Garry, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical School, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Lyubimov AV, Garry VF, Carlson RE, Barr DB, Baker SE. Simplified urinary immunoassay for 2,4-D: validation and exposure assessment. J Lab Clin Med. 2000 Aug;136(2):116-24. doi: 10.1067/mlc.2000.108150. PMID 10945240
- [Background] Lin N, Garry VF. In vitro studies of cellular and molecular developmental toxicity of adjuvants, herbicides, and fungicides commonly used in Red River Valley, Minnesota. J Toxicol Environ Health A. 2000 Jul 28;60(6):423-39. doi: 10.1080/00984100050033494. PMID 10933758
- [Background] Kirkhorn SR, Garry VF. Agricultural lung diseases. Environ Health Perspect. 2000 Aug;108 Suppl 4(Suppl 4):705-12. doi: 10.1289/ehp.00108s4705. PMID 10931789
- [Background] Garry VF, Burroughs B, Tarone R, Kesner JS. Herbicides and adjuvants: an evolving view. Toxicol Ind Health. 1999 Jan-Mar;15(1-2):159-67. doi: 10.1191/074823399678846619. PMID 10188198
- [Background] Schreinemachers DM, Creason JP, Garry VF. Cancer mortality in agricultural regions of Minnesota. Environ Health Perspect. 1999 Mar;107(3):205-11. doi: 10.1289/ehp.99107205. PMID 10064550